CLINICAL TRIAL: NCT00767650
Title: Neuropsychological Effects of Immunosuppressive Treatment in Subjects With Aplastic Anemia
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080222; 08-H-0222
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-28

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia; Cyclosporine; Campath; Neurophyschological Side Effect
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will use neuropsychological tests to look at nervous system side effects of Cyclosporine (CsA) in patients with aplastic anemia. CsA is used as part of an immunosuppressive regimen in treating severe aplastic anemia. The drug can produce nervous system side effects, such as tremor and, less commonly, insomnia, anxiety, headache, confusion or seizures. This study will look at effects of CsA on intellectual ability, depression, anxiety, attention, concentration, memory, perception, coordination, and thought processing in patients

Patients 15 years of age or older who have severe aplastic anemia may be eligible for this study if they:

* are co-enrolled in a Clinical Center protocol in which they will receive CsA
* have not taken CsA for 6 months before enrolling in this study

Participants undergo neuropsychological testing. In addition, they provide blood samples and their clinical data are reviewed for things that may influence the interpretation of findings from the testing, such as results of blood tests, types of medications taken, number of transfusions required, etc. The procedures are as follows:

Before first dose of cyclosporine:

* Patients are asked about prior problems with their nervous system, prior treatment for their aplastic anemia (including transfusions), prior infections, and current medications. They then complete the following sets of tests:
* Battery 1: A set of three tests that measure intellectual ability, level of depression (if any) and level of anxiety (if any).
* Battery 2: A set of seven tests that measure changes in the central nervous system and how these changes affect attention, concentration, memory, perception, coordination, and thought processing.
* Patients provide a half teaspoon of blood for this study at the same time blood is collected for their primary treatment protocol.

  6 months and 12 months after starting cyclosporine
* Patients are asked about treatment for their aplastic anemia (including transfusions), infections, and changes in medications that have occurred since they started taking cyclosporine. They then repeat the set of tests in Battery 2.
* Patients provide a half teaspoon of blood for this study at the same time blood is collected for their primary treatment protocol.

DETAILED DESCRIPTION:
Cyclosporine (CsA) is widely used in the treatment of aplastic anemia as well as to provide immunosuppression after transplantation. CsA has a spectrum of neurologic and more subtle, poorly investigated neuropsychological functional effects. In the NHLBI, a unique opportunity exists to evaluate changes in neuropsychological function following CsA in a large cohort of aplastic anemia patients accrued to NHLBI treatment protocols.

With increased success in treating blood diseases with immunosuppressive therapy or stem cell transplantation that utilize CsA in the treatment regimen, patients are enjoying prolonged survival during which quality of life becomes an increasingly relevant concern. We therefore propose this natural history protocol designed to evaluate neuropsychological functioning before, during, and after CsA administration in severe aplastic anemia patients.

The primary objective is to evaluate changes in attention, language, memory, spatial/motor and executive function domains following CsA therapy using well established neuropsychological tests including the Neuropsychological Assessment Battery (NAB) Screening Module, Revised Hopkins Verbal Learning Test, Revised Brief Visual-spatial Memory Test, Judgment of Line Orientation test, Grooved Pegboard, Trail Making Test and the two performance subsets in Wechsler Adult Intelligence Scale-III. IQ test by Wechsler Abbreviated Scale of Intelligence and depression/anxiety level will be screened once prior to formal testing. Measures will also be correlated with clinical status, standard CsA side effects, CsA drug levels and relevant biochemical lab values at each time point to control the testing accuracy and explore potential correlation.

ELIGIBILITY:
* INCULSION CRITERIA:
* Diagnosed with aplastic anemia.
* Co-enrolled on a Clinical Center CsA treatment protocol that prescribes CsA (included but not limited to initial treatment cohort in both rabbit and horse ATG arm for the aplastic anemia patients).
* Age greater than or equal to 15 years old.

EXCLUSION CRITERIA:

* Prior use of cyclosporine within 6 months to next line of treatment.
* History of learning disability (i.e. dyslexia).
* Unable to read and speak English (the neuropsychological testing tools are validated for use in English speaking subjects only).
* Life expectancy less than six months or when clinical status prevents full performance with testing.
* Either adult patients or guardians for the minor patient, unable to comprehend the investigational nature of the study and provide informed consent.
* Inability or unwillingness to come to Clinical Center for the 6-month and 12-month follow-up appointments.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-09-23; Study Completion 2011-06-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Gijtenbeek JM, van den Bent MJ, Vecht CJ. Cyclosporine neurotoxicity: a review. J Neurol. 1999 May;246(5):339-46. doi: 10.1007/s004150050360. PMID 10399863
- [Background] Syrjala KL, Dikmen S, Langer SL, Roth-Roemer S, Abrams JR. Neuropsychologic changes from before transplantation to 1 year in patients receiving myeloablative allogeneic hematopoietic cell transplant. Blood. 2004 Nov 15;104(10):3386-92. doi: 10.1182/blood-2004-03-1155. Epub 2004 Jul 13. PMID 15251983